CLINICAL TRIAL: NCT01589718
Title: A Phase III Randomized 1:1, Masked, Study of the Safety, Tolerability, and Efficacy of Intravitreal Pre-op 0.3mg Pegaptanib Sodium Versus Sham, for Adjuvant Management of TRD and Vit Hem Associated With PDR
Brief Title: A Study of the Safety, Tolerability, and Efficacy of IVT Pre-op 0.3mg Pegaptanib Sodium Versus Sham, for Management of Tractional Retinal Detachment and Vitreous Hemorrhage With Proliferative Diabetic Retinopathy
Acronym: No-Crunch01
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patients were enrolled
Sponsor: Greater Houston Retina Research (Other)
Responsible Party: Principal Investigator, James C. Major, PhD, MD, Principal Investigator, Greater Houston Retina Research
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: No-Crunch 01
Record Dates: First submitted 2012-04-27; First posted 2012-05-02 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative Diabetic Retinopathy; Tractional Retinal Detachment; Vitreous Hemorrhage
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — pegaptanib; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.3mg Pegaptanib Sodium, Macugen (Experimental): will receive Macugen intravitreal injection prior to surgery
  Interventions: Drug: Macugen
- Sham injection (Sham Comparator): will receive a sham injection
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: Macugen — one intravitreal injection of Macugen prior to vitrectomy surgery
  Other Names: 0.3mg Pegaptanib Sodium, Macugen
  Arms: 0.3mg Pegaptanib Sodium, Macugen
Drug: Sham — The subject in cohort 2 will receive one sham comparator, sham injection prior to vitreous surgery.
  Arms: Sham injection

SUMMARY:
The purpose of this study is to assess whether preoperative pegaptanib sodium safely improves vitreous hemorrhage prior to surgical intervention and to evaluate the stability of pre-existing tractional retinal detachment.

DETAILED DESCRIPTION:
Patients undergoing pars plana vitrectomy for active PDR with TRD will receive a single intravitreal pre-operative 0.3mg Macugen™ prior to surgery versus sham injection.

Specific timing of the injection will be at no sooner than 7 days and no longer than 14 days prior to surgery.

Patients will receive a preinjection fundus photo and another post injection photo the day of surgery as dictated by the operative schedule.

Some photos may be limited secondary to vitreous hemorrhage. Follow up visits after surgery will be one day, one week, one month, and three months.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity in the study eye between 20/30 and light perception (LP)
* Willingness to provide signed informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Age ≥ 18 years
* For sexually active women of childbearing potential, agreement to the use of an appropriate form of contraception (or abstinence) for the duration of the study

Exclusion Criteria:

* History of anti-VEGF treatment in the study eye
* History of previous pars plana vitrectomy in the study eye
* Intraocular surgery in the study eye within one month of the study
* Patients with extensive vitreous hemorrhage in conjunction with a rhegmatogenous retinal detachment
* Tractional retinal detachment from causes inconsistent with PDR, such as inflammation or trauma
* Any concurrent intraocular condition in the study eye that could either require medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition or if allowed to progress untreated could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA over the study period.
* Active intraocular inflammation (grade trace or above) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as IOP≥ 35 mmHg despite treatment with anti-glaucoma medication)
* History of glaucoma-filtering surgery in the study eye
* History of corneal transplant in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Tractional Retinal Detachment Repair | 6 months
  Overall score of perceived improvement during surgery as determined by a surgeon's subjective questionnaire.

SECONDARY OUTCOMES:
Post surgical interventions | 6 Months
  Post surgical interventions including need for additional surgery, additional injections or PRP laser
Vitreous Hemorrhage and Tractional Retinal Detachment Improvement | 6 months
  Pre and perioperative fundus photo comparisons on an objective scale
Adverse Events | 6 months
  Incidence and severity of ocular and nonocular adverse events, such as redetachment, progression to neovascular glaucoma, endophthalmitis, etc. through post operative month 3
Visual Acuity | 6 months
  Visual acuity as measured by BCVA

CONTACTS AND LOCATIONS:
Overall Officials: James C Major, MD, Principal Investigator — PI
Locations (1):
- Retina Consultants of Houston, Houston, Texas, United States

REFERENCES:
- [Background] Gonzalez VH, Giuliari GP, Banda RM, Guel DA. Intravitreal injection of pegaptanib sodium for proliferative diabetic retinopathy. Br J Ophthalmol. 2009 Nov;93(11):1474-8. doi: 10.1136/bjo.2008.155663. Epub 2009 Aug 18. PMID 19692371
- [Background] Wroblewski JJ, Wells JA 3rd, Gonzales CR. Pegaptanib sodium for macular edema secondary to branch retinal vein occlusion. Am J Ophthalmol. 2010 Jan;149(1):147-54. doi: 10.1016/j.ajo.2009.08.005. Epub 2009 Oct 28. PMID 19875087
- [Background] Chen E, Park CH. Use of intravitreal bevacizumab as a preoperative adjunct for tractional retinal detachment repair in severe proliferative diabetic retinopathy. Retina. 2006 Jul-Aug;26(6):699-700. doi: 10.1097/01.iae.0000225351.87205.69. No abstract available. PMID 16829817
- [Derived] Dervenis P, Dervenis N, Smith JM, Steel DH. Anti-vascular endothelial growth factors in combination with vitrectomy for complications of proliferative diabetic retinopathy. Cochrane Database Syst Rev. 2023 May 31;5(5):CD008214. doi: 10.1002/14651858.CD008214.pub4. PMID 37260074